CLINICAL TRIAL: NCT00382941
Title: Study of LED Phototherapy for Musculoligamentous Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hermano Miguel Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FT-01-05-05
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Tendinopathy; Sprains and Strains; Muscle Spasm; Epicondylitis; Fasciitis
MeSH Terms: conditions — Tendinopathy; Sprains and Strains; Spasm; Fasciitis

INTERVENTIONS:
Device: Red and near infrared LED phototherapy device

SUMMARY:
The purpose of this study is to determine whether LED phototherapy using combined red and near infrared light (approved: Ministry of Health of Russian Federation No. 29/06070997/1080-00, EUROCAT Certificate No. CP033321-IV) is effective in the treatment of musculoligamentous lesions in physiotherapy practice

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute or chronic musculoligamentous lesion
* Must be able to understand instructions and fill in auto administered questionnaires
* Informed consent

Exclusion Criteria:

* Use of oral corticosteroids or corticosteroid injections
* Systemic diseases
* General contraindications for phototherapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sergiy Voznesenskyy, PhD, BPT, Principal Investigator — Hermano Miguel Foundation
Locations (3):
- Ecuador (3):
  - CAID, Hermano Miguel Foundation, Quito, Pichincha
  - Health Service, UDV Quito Centro Occidente, National Police of Ecuador, Quito, Pichincha
  - Rehabilitation Department, A.B.E.I. Foundation, Quito, Pichincha